CLINICAL TRIAL: NCT01778491
Title: AMD Phenotype and Genotype Study (APGS)
Brief Title: AMD Phenotype and Genotype Study
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130027; 13-EI-0027
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-09-29

CONDITIONS: Age-Related Macular Degeneration; AMD
Keywords: Phenotype-Genotype correlation; Phenotype; Phenotypes; Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Age-related macular degeneration (AMD) is a disease that blurs the sharp vision needed for activities such as reading, sewing, and driving. It affects the macula, the center of the retina at the back of the eye, which allows a person to see fine detail. Researchers want to collect medical histories, eye exam data, and genetic information that may be associated with AMD. They want to compare this information with information collected from people without AMD.

Objectives:

- To collect medical information and gene samples for researchers studying AMD.

Eligibility:

* Individuals between and 60 and 90 years of age who have AMD in at least one eye.
* Individuals between and 60 and 90 years of age who have no AMD in either eye.

Design:

* This study will involve one study visit. This study visit will last 6 to 8 hours.
* Participants will have the following tests and exams as part of their study visit:
* Full physical exam and medical history
* Full eye examination
* Laser scan of the eye
* Retina function test
* Vision sensitivity test
* Optional blood sample (for genetic study)
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
Objective: Late age-related macular degeneration (AMD) is the leading cause of blindness among elderly in the United States. At present the current classification systems do not take into consideration advances in imaging technology and genotyping and phenotyping.

Clinical centers in the US and around the world will conduct a pilot cohort study that will bring together resources and commitment to test the feasibility of developing a new classification scheme for AMD using imaging and visual function biomarkers, with the potential of correlating genetic information obtained in the future. These data could eventually help develop an understanding of the mechanisms involved in the development and progression of AMD. A database of men and women with and without AMD will be established and maintained. The project will recruit participants who have various stages of AMD and controls. The pilot study will identify the feasibility of obtaining imaging and visual function data and help identify which of these modalities should be included in a full scale longitudinal study, as well as how frequently and at which sites they should be obtained. All data, images and any potential biospecimens from the full scale longitudinal study will be available to researchers worldwide to help in the development of biomarker identification and classification development. The initiative should provide an unparalleled state-of-the-art standardized phenotype/genotype including AMD status with information on imaging, visual function, and biospecimen biomarkers. This study is the first phase of this initiative to test the feasibility and logistics of defining a standard database including enhanced phenotype and genotype data.

Study Population: This cohort study will recruit a minimum of 200 total participants with various stages of AMD, including controls and obtain the appropriate images and measures of visual function needed for the investigation and validation of an AMD phenotype.

Design: This cohort study is a multi-national, multi-center, observational study focused on AMD. The study is a pilot to test the ability to create an archive of data, biological samples (collected at other study sites), measures of visual function and ophthalmic images collected over time from a very well clinically characterized population of participants with a diagnosis of AMD. The database will also include a control group consisting of participants without a diagnosis of AMD.

Outcome Measures: The design of this cohort study and the data being collected will allow users to assess phenotypes of AMD, develop and evaluate potential markers and risk factors, develop and evaluate an AMD classification scheme(s), and assess the progression of the disease and investigate factors that shape it. It is not practical to anticipate all of the potential uses of the data, or all the types of analyses that will be performed to address user-defined questions.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

-Male or female participants must fall into any of the following categories:

* No drusen or any AMD-associated pigment abnormalities (no apparent aging changes)
* Small drusen (less than or equal to 63 micro millimeters in diameter) and the absence of AMD-associated pigment abnormalities in either eye (normal aging changes)
* Medium (>63 (Micro)m and less than or equal to 125 micro millimeters in diameter) drusen in either eye (Early AMD)
* Large (>125 (Micro)m in diameter) drusen with or without pigmentary abnormalities in either eye (Intermediate AMD)
* Neovascular AMD in only one eye or the presence of geographic atrophy in either eye but with vision >20/60 in the better-seeing eye (Late AMD)
* Presence of reticular Drusen in either eye

AMD classification will be based on clinical evaluation.

* 60 years of age or older
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Retinal photographs of sufficient quality to allow assessment of the macular area for AMD lesions including drusen

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present:

* Presence of lens or vitreous opacity in eye(s) with AMD to preclude adequate ophthalmic imaging
* Presence of ocular conditions that may now or in the future complicate the evaluation of AMD [e.g., vascular occlusion, diabetic retinopathy (>4 microaneurysms), etc.] in the eye(s) with AMD
* High myopia -6 Diopters or more severe
* Diagnosis of nystagmus
* Glaucoma with definite visual field defects. Participants with a history of the diagnosis of glaucoma, past or present use of medications to control intraocular pressure, or disc/nerve fiber layer defects suggestive of glaucoma can be eligible for the study if they have a documented normal Goldmann, Humphrey, or Octopus perimetry test within 6 months prior to qualification.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2012-11-05; Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
Allow users to assess phenotypes of AMD | 5 years
Develop and evaluate potential markers and risk | 5 years
Develop and evaluate an AMD classification scheme(s) | 5 years
Assess the progression of the disease and investigate that shape it. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- University of Bonn, Bonn, Germany

REFERENCES:
- [Background] Kini MM, Leibowitz HM, Colton T, Nickerson RJ, Ganley J, Dawber TR. Prevalence of senile cataract, diabetic retinopathy, senile macular degeneration, and open-angle glaucoma in the Framingham eye study. Am J Ophthalmol. 1978 Jan;85(1):28-34. doi: 10.1016/s0002-9394(14)76661-9. PMID 619683
- [Background] Smiddy WE, Fine SL. Prognosis of patients with bilateral macular drusen. Ophthalmology. 1984 Mar;91(3):271-7. doi: 10.1016/s0161-6420(84)34309-3. PMID 6201789